CLINICAL TRIAL: NCT02305628
Title: Post-Marketing Surveillance of Herceptin Subcutaneous in Breast Cancer
Brief Title: An Observational Study of Herceptin SC Safety in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29625
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort: Method of continuous surveillance per standard of care

SUMMARY:
This is a phase IV, prospective, multicenter, observational study (regulatory post-marketing surveillance) in approximately 600 patients who are to receive Herceptin SC (trastuzumab, subcutaneous administration) per approved local labeling. Patients will be under observation according to standard of care in Korea.

ELIGIBILITY:
Inclusion Criteria:

- All patients administered Herceptin SC for the locally approved indications

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment for breast cancer with Herceptin SC under observation according to standard of care and in line with the current local labeling in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-06-26 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Safety (composite outcome measure): Incidence of adverse events (AEs), serious adverse events (SAEs), adverse events of special interest, pregnancies, adverse drug reactions (ADRs); unexpected ADRs; expected ADRs | Up to 6 years

SECONDARY OUTCOMES:
Efficacy: Pathological Complete Response (pCR) in neoadjuvant early breast cancer (EBC) | Up to 6 years
Efficacy: Overall response per Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- South Korea (23):
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Myongji Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Ajou University Medical Center, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Gyeongsang National University Hospital, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Wonkwang University School of Medicine & Hospital, Jeonlabuk-do
  - Samsung Medical Center, Seoul
  - Inje University, Sanggye-Paik Hospital, Seoul
  - Korea Cancer Hospital of Korea Institute of Radiological and Medical Sciences, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Cheil General Hospital & Women's Healthcare Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - Borame Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Miz Medi Hospital, Seoul
  - Ulsan University Hosiptal, Ulsan